CLINICAL TRIAL: NCT00703443
Title: The Genetics of Cardiomyopathy and Heart Failure
Status: Withdrawn | Type: Observational
Why Stopped: Non applicable clinical trial
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: HS# 2007-5577; NIH/NHLBI 5K08HL081222-02
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Dilated Cardiomyopathy; Hypertrophic Cardiomyopathy; Mitochondrial Cardiomyopathy; Noncompaction Cardiomyopathy; Restrictive Cardiomyopathy
Keywords: Genetics; Dilated Cardiomyopathy; Hypertrophic Cardiomyopathy; Mitochondrial Cardiomyopathy; Noncompaction Cardiomyopathy; Restrictive Cardiomyopathy; Heart Failure
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Cardiomyopathy, Restrictive; Heart Failure

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood, Saliva, Buccal cells
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the genetic basis of cardiomyopathies and heart failure.

DETAILED DESCRIPTION:
The purpose of this research study is to explore the causes and inheritances of cardiomyopathies. Cardiomyopathies are serious medical conditions that result in a wide range of cardiac problems, from no symptoms at all to heart failure. The underlying genetics of cardiomyopathies are poorly understood. This study will collect personal, family, and medical history information to create a database of participants with cardiomyopathies. This information will be used to identify inheritance patterns within families with cardiomyopathies. In addition, samples from participants will be studied in the lab to see if any changes in their genetic information can be identified that would cause a cardiomyopathy. Overall, the research study is aimed at determining the cause of these cardiac conditions so that tests and treatments might be developed in the future.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a diagnosis of cardiomyopathy
* Family members of individuals with a diagnosis of cardiomyopathy
* Individuals with a nuclear mutation shown to confer risk of cardiomyopathy but who do not themselves have cardiomyopathy

Exclusion Criteria:

* Individuals who do not have cardiomyopathy, a relative with cardiomyopathy, or a nuclear mutation predisposing to cardiomyopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We are recruiting both local participants (who have been evaluated at UCI) and remote participants (who have been referred from outside UCI) with familial and simplex cases of hypertrophic, dilated, noncompaction, restrictive, and mitochondrial cardiomyopathies. As a control group, we are also recruiting patients with nuclear mutations known to increase the risk of cardiomyopathy, but who have not themselves developed cardiomyopathy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Zaragoza, M.D., Ph.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

REFERENCES:
- [Background] Zaragoza MV, Arbustini E, Narula J. Noncompaction of the left ventricle: primary cardiomyopathy with an elusive genetic etiology. Curr Opin Pediatr. 2007 Dec;19(6):619-27. doi: 10.1097/MOP.0b013e3282f1ecbc. PMID 18025927